CLINICAL TRIAL: NCT00620711
Title: IRB# 070984 "Pilot Study of Head Cooling in Preterm Infants With Hypoxic Ischemic Encephalopathy"
Brief Title: Pilot Study of Head Cooling in Preterm Infants With Hypoxic Ischemic Encephalopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, William Walsh, Professor of Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070984
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic ischemic encephalopathy; HIE; Neonatal encephalopathy; Cooling; hypothermia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Babies that meet criteria will be offered participation in feasibility trial, there are no other arms.
  Interventions: Device: Olympic Cool Cap

INTERVENTIONS:
Device: Olympic Cool Cap — Olympic Cool Cap will be applied to infants 32-35 weeks gestation who meet criteria for HIE.
  Other Names: Selective Head Cooling

SUMMARY:
The hypothesis is that premature infants' can have enough cooling applied to cool their brain to decrease CNS injury without cooling their body.

DETAILED DESCRIPTION:
Hypoxic ischemic encephalopathy (HIE) is a potentially devastating disease of the newborn central nervous system (CNS) . Portions of the CNS are deprived of oxygen and blood flow for a period of time which may lead to permanent brain injury manifested as cerebral palsy as well as cognitive defects. Until recently no treatment has been shown to be effective for preventing brain damage, even though it has been demonstrated that the damage is progressive and that there is a window of opportunity to arrest some of the evolving brain injury. However, in May of 2007 the FDA approved the first device specifically designed to ameliorate brain damage in term babies with HIE. This head cooling device which was studied here at Vanderbilt under IRB protocol 990129 Brain Cooling for the treatment of perinatal hypoxic ischemic encephalopathy. We thus have eight years of experience of using this device in term infants. The results of the initial trial demonstrated a successful reduction of HIE induced brain injury from 66% in control infants to 55% in treated babies. There were no significant risks to the application of this device in term babies who are kept cool for 72 hours after experiencing an acute HIE event. The initial trials were limited to term babies because of concern that premature infants would be more at risk for hypothermia induced problems such as hypoglycemia,and coagulopathy. The concern about hypothermia in preterm infants remains a limiting consideration for doing whole body cooling in this population. We propose to apply the cooling cap to the heads of preterm infants who have experienced a significant HIE injury but maintain their body temperature in the normal range (36.1-37° C rectally). Infants will be cooled for up to 72 hours and will be tracked till discharge. Although this is a feasibility study, the participants will also be followed-up at 6, 12 and 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Babies < 36 weeks gestation but > 32 0/7 weeks. These babies should be small enough to allow brain cooling with water circulating in a cooling cap applied to the surface of their head
* At least one of the following four criteria which are standard definitions for HIE:

  * Apgar 0-3 at 1,5,10 minutes due to hypoxia
  * pH less than 7.0
  * Base deficit greater than 15
  * Need for continued resuscitation due to hypoxia at 10 minutes
* AND a physical exam with evidence of hypotonia or lethargy or seizures indicative of evolving HIE.
* Intubated
* Age less than 6 hours
* Signed informed consent by parent / legal guardian
* Previous participant has been followed through 7 day head ultrasound.

Exclusion Criteria:

* Mild HIE will not be cooled, therefore babies without hypotonia or lethargy and babies who are not intubated will be excluded.
* Gestational age ≥ 36 weeks or < 32 weeks or less than 1200 grams.
* Older than 6 hours of age
* Infant deemed in extremis on clinical exam.
* Survival not expected, i.e. received 3 intravenous doses of epinephrine or more during resuscitation; on infusion of dopamine, dobutamine and/or epinephrine at time of evaluation; and/or has fixed/dilated pupils.
* Evidence of head trauma or skull fracture causing major intracranial hemorrhage
* Intraventricular hemorrhage
* Weight less than the 5th percentile for gestational age
* Refusal of consent
* Imperforate anus

Ages: 30 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2008-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willaim F Walsh, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Monroe Carell Jr Children's Hospital, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Shankaran S. Outcomes of hypoxic-ischemic encephalopathy in neonates treated with hypothermia. Clin Perinatol. 2014 Mar;41(1):149-59. doi: 10.1016/j.clp.2013.10.008. PMID 24524452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Preterm Infants meeting criteria for HIE 6 hours old
Groups:
- Group 1 Cool- Cap Applied While Maintaining Rectal Temp: Babies that meet criteria will be offered participation in feasibility trial, there are no other arms.
Period: Overall Study
Arm/Group | Group 1 Cool- Cap Applied While Maintaining Rectal Temp
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Preterm infants with HIE
Groups:
- Preter Infnats With HIE: Babies that meet criteria will be offered participation in feasibility trial, there are no other arms. Criteria include Sentinel evnet , Low Apgar, pH less than 7, Neonatal encephalopathy with no other cause and need for mechanical ventialtion
  Olympic Cool Cap: Olympic Cool Cap will be applied to infants 32-35 weeks gestation who meet criteria for HIE.
Arm/Group | Preter Infnats With HIE
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Trial- the Olympic Cool Cap Will be Applied, Can the Delivered Cap Temperature be Less Than 12 Degrees Without Changing Rectal Temperature.
Description: Measurement of number of participants able to obtain 12 degree cap temperature
Time Frame: 60 minutes intervals up to 72 hours
Population: all analysized
Measure: Number; unit: participants
Arm/Group | Group 1 Cool- Cap Applied While Maintaining Rectal Temp
Number analyzed (Participants) | 4
participants | 2

2. Primary Outcome: Cap Cooled to 12 Degrees Without Reducing Rectal Temperature
Description: Yes/no
Time Frame: 6 hours
Measure: Number; unit: participants
Arm/Group | Group 1 Cool- Cap Applied While Maintaining Rectal Temp
Number analyzed (Participants) | 4
participants | 2

ADVERSE EVENTS:
Groups:
- Preterm Infants With HIE: Babies that meet criteria will be offered participation in feasibility trial, there are no other arms.
  Olympic Cool Cap: Olympic Cool Cap will be applied to infants 32-35 weeks gestation who meet criteria for HIE.
Arm/Group | Preterm Infants With HIE
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preterm Infants With HIE (N=4)
Death (General disorders) | 1 (2) — Family withdrew patient due to poor prognosis
Intracranial Hemorrhage (Nervous system disorders) | 1 (1) — Intracranial hemorrhage

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes